CLINICAL TRIAL: NCT06242665
Title: You Are What You Eat: Food As a Risk Factor and a Treatment for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Ashley Gearhardt, Professor of Psychology, College of Literature, Science, and the Arts, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HUM00231527
Record Dates: First submitted 2024-01-16; First posted 2024-02-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-08

CONDITIONS: Depression
Keywords: Depression; Blood Glucose; Ultra-Processed Foods
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Multi-method, mixed-design
Who Masked: Participant
Masking Description: Participants will be blinded to their condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meal Delivery (Experimental): Dietary change (low ultra-processed meal delivery) and nutrition guidance to follow a low UPF diet.
  All participants complete a series of three in-lab visits with remote data collection:
  Visit 1 and the following week comprise the baseline assessment period.
  Visit 2 and the following 2 weeks comprise the dietary intervention period. Meal delivery and nutritional guidance is provided by the study team for 14 days in accordance with a low UPF diet.
  Visit 3 comprises post-intervention assessment All participants will complete remote assessments at 1 month and 6 month follow-ups.
  Interventions: Other: Low UPF Meals (Study Provided); Other: Low UPF Nutritional Guidance
- Nutritional Guidance (Experimental): Dietary change (nutritional guidance)
  Visit 1 and the following week comprise the baseline assessment period.
  Visit 2 and the following week comprise the dietary intervention period. Nutritional guidance is provided by the study team for 14 days in accordance with a low UPF diet. Participants are delivered a box of snacks consistent with a low UPF diet.
  Visit 3 comprises post-intervention assessment. All participants will complete remote assessments at 1 month and 6 month follow ups.
  Interventions: Other: Low UPF Nutritional Guidance; Other: Low UPF Snacks (Study Provided)

INTERVENTIONS:
Other: Low UPF Meals (Study Provided) — Meals provided through delivery service
  Arms: Meal Delivery
Other: Low UPF Nutritional Guidance — Self-guided instructions from study team.
Other: Low UPF Snacks (Study Provided) — Low UPF snacks provided to participant
  Arms: Nutritional Guidance

SUMMARY:
This study experimentally investigates 1) whether ultra processed food (UPF) intake contributes to depression by increasing low mood and poor sleep due to blood glucose fluctuations (which then increases the desire to consume more UPFs) and 2) to investigate the effectiveness of a 2-week meal-kit intervention that provides convenient and tasty minimally processed foods (MPF) to reduce depression. The following aims and hypotheses are tested:

Aim 1: To investigate whether UPF intake and low mood contribute to each other in a cyclical fashion through the mechanisms of blood glucose fluctuations and disrupted sleep in individuals with moderate-to-severe depression.

H1: It is hypothesized that UPF intake and high blood glucose will be associated with low mood in individuals with depression.

Aim 2: To establish an industry partnership to investigate whether commercially available meal kit delivery reduces symptoms of depression in individuals with moderate-to-severe depression relative to a nutrition education control condition.

H2: Meal kit delivery will lead to reductions in depression symptoms and daily reductions in low mood relative to the control condition (nutrition guidance only).

DETAILED DESCRIPTION:
The study will include a combination of in-person, at-home, and virtual activities over the course of ~21 days (contingent on scheduling, this duration may vary and particularly between in-person visits #1 and #2). Participants complete three in-lab visits, each followed by a week of remote data tasks (e.g., ecological momentary assessment, continuous glucose monitoring, and physical activity and sleep tracking (Fitbit)).

During in-lab visit #1, participants will complete questionnaires and interviews, have a continuous glucose monitor inserted, and will have body composition measurements taken (height, weight, Inbody scan). Participants will complete the remote tasks for the following week while eating their typical diet (i.e., baseline period).

During in-lab visit #2, participants will complete questionnaires, interviews, and body composition measurements (height, weight, Inbody scan). Participants are randomly assigned to a meal delivery (will receive two weeks of low UPF meals and nutrition guidance) or control (will receive some snacks and nutrition guidance) condition (i.e., dietary intervention period). Participants will complete the remote tasks for the following two weeks.

During in-lab visit #3, participants will complete questionnaires, interviews, and body composition measurements (height, weight, InBody scan).

Participants are contacted 1- and 6-months later to complete a short follow-up survey and provide information about their current diet.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Must own an Android or iPhone smartphone
* Must be able to access phone one every 90 minutes
* Able to attend consent call over zoom or phone
* Endorsement of a PHQ-8 score of at least 10 assessed at consent
* Endorsement of a PHQ-8 score of at least 8 assessed 24 hours prior to Visit 1
* Endorse daily intake of at least UPF foods
* Willing to come to three in-lab visits
* Willing to follow dietary guidelines
* Must be able to speak, write, and read English fluently

Exclusion Criteria:

* Regular smoking of cigarettes or vaping of nicotine
* History of medication that impact reward, eating, or indicate severe mental health conditions (e.g., Lithium)
* The following medical conditions; Diabetes Type I, Diabetes Type II, Prediabetes, Bipolar Disorder, Schizophrenia, Psychotic Disorder, Depression with psychotic symptoms, Borderline Personality Disorder, Hypoglycemia, Substance use disorder (e.g., alcohol use disorder, opioid use disorder, cannabis use disorder), Obsessive compulsive disorder, and Post-traumatic stress disorder
* Endorsement of a suicide attempt or having been hospitalized for psychiatric reasons in the last year
* A diagnosis of a restrictive eating disorder (anorexia nervosa, bulimia nervosa, purging disorder) within the last 5 years
* History of disorders that impact eating (e.g., cancer, irritable bowel syndrome, inflammatory bowel disease, hypothyroidism).
* Current pregnancy, breast-feeding, trying to get pregnant, or within six months of having given birth
* Frequent (i.e., weekly) night shift work or irregular shifts and for abnormal sleep patterns (i.e., wake up time after 11am)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-12-09 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Low mood symptoms | Assessed during dietary adherence period for 2 weeks
  Depression symptoms (e.g., anhedonia, low energy) will be assessed with the Patient Health Questionnaire (PHQ-8) using ecological momentary assessment and at each study visit. The PHQ-8 scores 8 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Higher PHQ-8 scores indicate greater depression symptoms.

SECONDARY OUTCOMES:
Blood Glucose Level | Assessed during dietary adherence period for 2 weeks
  Assessed using a continuous blood glucose monitor
Sleep Quality | Assessed during dietary adherence period for 2 weeks
  Assessed using a Fitbit
Metabolic Equivalent of Task (METs) | Assessed during dietary adherence period for 2 weeks
  A measure of physical activity engagement assessed using a Fitbit
Feasibility of the Interventions | Assessed post-dietary change during in-lab Visit 3 (1 day)
  Assessed in a qualitative interview at Visit 3
Accessibility of the Interventions | Assessed post-dietary change during in-lab Visit 3 (1 day)
  Assessed in a qualitative interview at Visit 3

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
This research will generate demographic, heart rate, ecological momentary assessment, continuous glucose monitoring, self-report and anthropometric data. The data will be stored as SPSS or SAS files. Meta data will also be included in the selected repositories. The metadata will include the data dictionaries, which describe the generation of all variables. The deidentified data will be made available within one year of completion of the study at the University of Michigan's data repository - Deep Blue.
Time Frame: Beginning 1 year and ending 7 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal will be able to access data to achieve aims outlined in the approved proposal. Proposals should be directed to agearhar@umich.edu to gain access. Data requestors will need to sign a data access agreement.